CLINICAL TRIAL: NCT05437055
Title: THUNDER: Acute Ischemic Stroke Study with the Penumbra System® Including Thunderbolt™ Aspiration Tubing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21340
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion
Keywords: Acute Ischemic Stroke; AIS; Large Vessel Occlusion; LVO; Mechanical Thrombectomy; Penumbra System; Thunderbolt Aspiration Tubing; A Direct Aspiration First Pass Technique; ADAPT
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): Use of Penumbra System including Thunderbolt in patients with acute ischemic stroke secondary to intracranial large vessel occlusion who are eligible for mechanical thrombectomy
  Interventions: Device: Mechanical Thrombectomy (Penumbra System with Thunderbolt)

INTERVENTIONS:
Device: Mechanical Thrombectomy (Penumbra System with Thunderbolt) — Subject will receive Penumbra System with Thunderbolt

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of the Penumbra System including Thunderbolt Aspiration Tubing (Thunderbolt) in a population presenting with acute ischemic stroke (AIS) secondary to intracranial large vessel occlusion (LVO) who are eligible for mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 - 80 years
2. Treatment within 8 hours of symptom onset
3. Pre-stroke mRS 0-2
4. Patient experiencing acute ischemic stroke secondary to intracranial large vessel occlusion in the internal carotid, middle cerebral (M1 or M2), basilar, or vertebral artery
5. If patient is eligible for thrombolytic therapy, it was administered as soon as possible, and no later than 3 hours from stroke symptom onset
6. Planned frontline treatment with Penumbra System including Thunderbolt modulated aspiration
7. Informed consent obtained per Institution Review Board/Ethics Committee requirements

Exclusion Criteria:

1. Stenosis, excessive tortuosity, or any occlusion in a proximal vessel requiring treatment or preventing access to the thrombus
2. Alberta Stroke Program Early CT Score (ASPECTS) ≤6 or core infarct volume >50 mL on MRI or CT-based imaging (for anterior circulation strokes)
3. Pregnant patient
4. Life expectancy < 90 days due to comorbidities
5. Current participation in an interventional drug or device study that may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies
6. Other medical, behavioral, or psychological conditions that in the opinion of the Investigator could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Efficacy Endpoint: Angiographic Revascularization | Immediate Post Procedure
  Angiographic revascularization of the occluded target vessel at immediate post-procedure as defined by mTICI 2b or higher.
  *mTICI ranges from 0-3, with higher grading representing better outcome

SECONDARY OUTCOMES:
Efficacy Endpoint: Angiographic Revascularization After First Pass | Index Procedure
  Angiographic revascularization of the occluded target vessel after first pass as defined by mTICI 2b or higher
  *mTICI ranges from 0-3, with higher grading representing better outcome
Efficacy Endpoint: Angiographic Revascularization | Immediate Post Procedure
  Angiographic revascularization of the occluded target vessel at immediate post-procedure as defined by mTICI 2c or higher
  *mTICI ranges from 0-3, with higher grading representing better outcome
Efficacy Endpoint: Time to Revascularization | Index Procedure
  Time to Revascularization
Efficacy Endpoint: Modified Rankin Scale (mRS) | 90 Days Post-Procedure
  Functional outcomes measured by mRS 0-2 at 90 days
  (0 no symptoms - 5 severe disability)
Safety Endpoint: Rate of Symptomatic Intracranial Hemorrhage (sICH) | 24 hours Post-Procedure
  Occurrence of symptomatic intracranial hemorrhages (sICH) at 24 hours
Safety Endpoint: All-cause mortality | 90 Days Post-Procedure
  All-cause mortality at 90 days
Safety Endpoint: Serious Adverse Events (SAEs) | Up to 24 hours Post-Procedure
  Incidence of device related, and/or procedure related Serious Adverse Events (SAEs) within 24 hours post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Donald Frei, M.D., Principal Investigator — HCA HealthONE, LLC (Swedish Medical Center); David Fiorella, M.D., Principal Investigator — The Research Foundation for The State University of New York (Stony Brook University)
Locations (32):
- United States (32):
  - Abrazo West Campus, Goodyear, Arizona
  - Sharp Grossmont, San Diego, California
  - HRI - Swedish, Englewood, Colorado
  - Yale New Haven, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - Jackson Memorial (U. of Miami), Miami, Florida
  - St. Joseph - BayCare, Tampa, Florida
  - Piedmont Hospital Atlanta, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - North Shore U., Evanston, Illinois
  - Edward Elmhurst Health, Naperville, Illinois
  - Indiana U. Health, Indianapolis, Indiana
  - KUMC, Kansas City, Kansas
  - Massachusetts General, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Abbott Northwestern, Minneapolis, Minnesota
  - St. Dominic, Jackson, Mississippi
  - Nebraska Medical, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Stonybrook U., Stony Brook, New York
  - New Hanover Regional, Wilmington, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Wellspan York, York, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Fort Sanders, Knoxville, Tennessee
  - Methodist U., Memphis, Tennessee
  - UT Houston, Houston, Texas
  - Christus Trinity Medical Center, Tyler, Texas
  - Riverside Regional Medical Center, Newport News, Virginia
  - Valley Medical Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No